CLINICAL TRIAL: NCT01272141
Title: Phase II Trial of Lapatinib in Combination With Everolimus in Triple Negative Metastatic or Locally Advanced Breast Cancer
Brief Title: A Study of Lapatinib in Combination With Everolimus in Patients With Advanced, Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, Funding stopped
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Read, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00031112; WCI1711-09 (Other: Other)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Breast Neoplasms; Breast Cancer; Cancer of the Breast
Keywords: Metastatic breast cancer; Triple negative breast cancer; Estrogen receptor (ER)/progesterone receptor (PR)/human epidermal growth factor receptor 2 (HER2)-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Lapatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A: Lapatinib plus Everolimus (Experimental)
  Interventions: Drug: Lapatinib and Everolimus

INTERVENTIONS:
Drug: Lapatinib and Everolimus — Lapatinib: 1250 mg by mouth daily
  Everolimus: 5mg by mouth daily
  Other Names: Lapatinib; Tykerb; Everolimus; Affinitor

SUMMARY:
The patient is being asked to join this clinical research study to find out if lapatinib, an agent that targets a protein, called epidermal growth factor receptor (EGFR) on the surface of cancer cells in combination with everolimus, an agent that targets a protein in the cancer cell, called mammalian target of rapamycin (mTOR) is effective in metastatic triple negative breast cancers that are no longer controlled by standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ER(-), PR(-), HER2(-) locally advanced or metastatic breast cancer
* Disease progression following prior first line cytotoxic chemotherapy in metastatic setting
* At least 1 lesion measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Age >18 years old
* Female
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Left ventricular ejection fraction (LVEF) > 50%
* Absolute neutrophil count (ANC)>1500/mm3; platelets >100,000/mm3; hemoglobin > 9 g/dL; serum creatinine < 1.5x upper limit of normal (ULN); total bilirubin < 1.5x ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN
* Patients must be recovered from both acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Patients of childbearing potential agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method)

Exclusion Criteria:

* Patients with current active hepatic or biliary disease (except for patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Patients with an active infection or with a fever > 101.3 Fahrenheit within 3 days of the first scheduled day of protocol treatment
* Patients with active central nervous system (CNS) metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for 3 weeks are eligible for the trial
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin or cervical intra-epithelial neoplasia with two consecutive normal pap smears 6 months apart
* Patients who received radiotherapy to more than 25% of their bone marrow; or patients who received radiotherapy to target lesions within 4 weeks of entry
* Patients who are receiving concurrent investigational therapy
* Peripheral neuropathy >= Grade 2
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of allogeneic transplant
* Known HIV or Hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Read, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Midtown (Crawford Long Hospital), Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Lapatinib Plus Everolimus
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A: Lapatinib Plus Everolimus
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  41-45 years | 2
  46-50 years | 2
  51-55 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Will Measured Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria. Tumor Assessment for All Lesions Must be Performed Every Eight Weeks While on Study by CT Scan.
Time Frame: Tumor assessment for all lesions must be performed by CT scan every 8 weeks while on study.
Population: No data were collected due to early termination.
Arm/Group | Arm A: Lapatinib Plus Everolimus
Number analyzed (Participants) | 0

2. Primary Outcome: The Safety and Toxicity of the Combination Therapy of Lapatinib and Everolimus Will be Monitored Using the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v. 3.0. The Incidence of Any Grade 3 or 4 Toxicities Will be Analyzed.
Time Frame: Safety assessments will be performed every four weeks while the patient remains on study.
Population: No data were collected due to early termination.
Arm/Group | Arm A: Lapatinib Plus Everolimus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm A: Lapatinib Plus Everolimus
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Lapatinib Plus Everolimus (N=5)
Shortness of breath due to pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes